CLINICAL TRIAL: NCT04789954
Title: An Exploratory Study to Evaluate the Dose Response-Relationship of Pharmacodynamic Parameters of AryoSeven, in Patients With Hemophilia With Inhibitors
Brief Title: Study on the Dose-response Relationship of Pharmacodynamic Parameters in Patients With Hemophilia With Inhibitors
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGA 2020-01
Record Dates: First submitted 2021-03-04; First posted 2021-03-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Hemophilia A With Inhibitor; Hemophilia B With Inhibitor
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AryoSeven 10 μg/kg (Experimental): Single dose, intravenously
  Interventions: Biological: Eptacog alfa, activated
- AryoSeven 30 μg/kg (Experimental): Single dose, intravenously
  Interventions: Biological: Eptacog alfa, activated
- AryoSeven 90 μg/kg (Experimental): Single dose, intravenously
  Interventions: Biological: Eptacog alfa, activated
- AryoSeven 270 μg/kg (Experimental): Single dose, intravenously
  Interventions: Biological: Eptacog alfa, activated
- NovoSeven 30 μg/kg (Active Comparator): Single dose, intravenously
  Interventions: Biological: Eptacog alfa, activated

INTERVENTIONS:
Biological: Eptacog alfa, activated — A dose sequence for each injection will be randomly selected from the following doses: 10 μg/kg, 30 μg/kg, 90 μg/kg, or 270 μg/kg, separated by a wash-out period of 3 days.

SUMMARY:
Randomized, double-blind, single-dose, 5 ways crossover, exploratory clinical trial evaluating four different doses of AryoSeven (eptacog alfa, activated) and NovoSeven on selected pharmacodynamic parameters in patients with hemophilia with inhibitors.

DETAILED DESCRIPTION:
Randomized, double-blind, single dose, 5 ways crossover, clinical trial evaluating four different doses (10 µg/kg, 30 µg/kg, 90 µg/kg, and 270 µg/kg) of AryoSeven (recombinant human FVII activated or eptacog alfa, activated) and one dose of NovoSeven (30 µg/kg) on selected pharmacodynamic parameters (PD) [Primary: Thrombin Generation Assay (TGA)] in male adult and adolescent (>12 years) patients with hemophilia A or B, with an inhibitors titer >5 Bethesda Units [BU] and not in bleeding status. This will be an exploratory study to evaluate dose-response relationship of PD markers as surrogate efficacy endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital haemophilia A or B with inhibitors to FVIII or FIX titer >5 Bethesda Units [BU]
* with > 2 episodes of bleeding/year requiring treatment with FVII infusions, not in bleeding episode
* Male adults and adolescents (>12 years)
* Patient informed consent has been obtained [Patients to be enrolled must also provide voluntary written informed consent to the protocol prior to screening to be eligible for the study. For adolescents, parent/legal guardian must provide consent and, wherever possible, patient assent will also be obtained. For compromised patients, their designated proxy must provide informed consent].
* Patients willing and able to be hospitalized prior to time of study medication administration for plasma sampling (5 times during the study).

Exclusion Criteria:

* Any other type of congenital or acquired coagulopathy, such as: liver disease (hepatitis), vitamin k deficiency, uremia, malignancy.
* Antibodies against Factor VII
* Ongoing bleeding prophylaxis regimens with AryoSeven/NovoSeven or planned to occur during the trial
* Platelet count less than 100.000 platelets/mcL (at screening visit)
* Any clinical sign or known history of arterial thrombotic event or deep venous- thrombosis or pulmonary embolism
* HIV positive with current CD4+ count of less than 200/µL
* Liver cirrhosis
* Factor VIII/IX immune tolerance induction regimen planned to occur during the trial
* Known hypersensitivity to the study medication
* Parallel participation in another experimental drug trial.
* Parallel participation in another marketed drug trial that may affect the primary end-point of the study.
* Concomitant diseases and/or medications, or any other conditions, that render the patient unsuitable for inclusion into the study in the judgement of the investigator.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Lag time of the thrombin generation curve | Up to 30 hours after AryoSeven and NovoSeven injection
  Time to 16.7% of peak plasmatic concentration, in minutes.

SECONDARY OUTCOMES:
Endogenous Thrombin Potential (PD parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Area under the curve plasma levels of thrombin generation curve (in nmol/per minute)
Time to Peak (PD parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Time to Peak of thrombin generation curve (in minutes)
Peak height (PD parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Peak height of thrombin generation curve (in nmol/ml)
F1.2 prothrombin fragments (PD parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Peak height (micg/L)
D-dimer (PD parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Peak height (micg/L)
AUCinf (PK parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Area under the plasma concentration time curve from time 0 to infinity, based on the last observed concentration;
Cmax (PK parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Observed maximum plasma concentration
Time of Cmax (PK parameter) | Up to 30 hours after AryoSeven and NovoSeven injection
  Time of observed maximum plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Iacobelli, MD, Study Director — Consultant
Locations (1):
- Comprehensive Hemophilia Care Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No